CLINICAL TRIAL: NCT07197138
Title: Pilot Study on the Effects of Intensified Repetitive Transcranial Magnetic Stimulation on Immunological Blood Parameters in Patients With Depression and Comorbid Post-COVID-19 Condition
Brief Title: IMPACT-D+: Immune-Modulating and Psychometric Effects of Accelerated TMS in Depression Plus Comorbid Post-COVID-19 Condition
Acronym: IMPACT-D+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-0648
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder; Post-Acute COVID-19 Syndrome
Keywords: Major depressive disorder; Post-COVID-19-condition; neuropsychology; psychometry; Immunemarkers; IL-6; TNF; CRP; repetitive transcranial magnetic stimulation; intermittent theta burst; accelerated rTMS; neuroinflammation
MeSH Terms: conditions — Depressive Disorder; Post-Acute COVID-19 Syndrome; Depressive Disorder, Major; Neuroinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: Two active iTBS schedules: once-daily for 6 weeks vs six times daily for 5 days; total 30 sessions per participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard iTBS (once daily) (Active Comparator): Standard: Participants receive one iTBS session per day, Monday through Friday, for 6 weeks (total 30 sessions). Each session consists of intermittent theta-burst stimulation (iTBS) applied to the left dorsolateral prefrontal cortex (DLPFC) at 90% of resting motor threshold using a PowerMAG 100 ppTMS stimulator. Each session lasts approximately 3 minutes.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS) using PowerMAG 100 ppTMS
- Intensified iTBS (6x daily) (Experimental): Intensified: Participants receive six iTBS sessions per day at intervals of about 60 minutes, for 5 consecutive days (total 30 sessions). Each session uses the same iTBS parameters as in the standard arm: stimulation of the left dorsolateral prefrontal cortex (DLPFC) at 90% of resting motor threshold with a PowerMAG 100 ppTMS stimulator, lasting about 3 minutes per session.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS) using PowerMAG 100 ppTMS

INTERVENTIONS:
Device: Intermittent theta-burst stimulation (iTBS) using PowerMAG 100 ppTMS — iTBS at 90% resting motor threshold; bursts of 3 pulses at 50 Hz repeated at 5 Hz; ~3 minutes per session; applied to left dorsolateral prefrontal cortex; 30 total sessions; schedule per arm as specified.

SUMMARY:
This is a monocentric, randomized pilot study conducted at the Max Planck Institute of Psychiatry, Munich. The study investigates the effects of two different intermittent theta-burst stimulation (iTBS) schedules on biological and clinical outcomes in patients with depression and comorbid Post-COVID-19 condition (PCC). Participants will be randomized into two arms, both receiving a total of 30 active iTBS sessions applied to the left dorsolateral prefrontal cortex (DLPFC) at 90% resting motor threshold using a PowerMAG 100 ppTMS stimulator:

* Standard Arm: One iTBS session per day, five days per week, over six weeks.
* Intensified Arm: Six iTBS sessions per day, approximately one-hour apart, over five consecutive days.

The primary outcomes are changes in immunological blood markers (C-reactive protein [CRP], tumor necrosis factor [TNF], interleukin-1β [IL-1β], interleukin-6 [IL-6]) and depressive symptomatology measured by Beck Depression Inventory-II (BDI-II) and Montgomery-Asberg Depression Rating Scale (MADRS). Secondary outcomes include fatigue (Fatigue Severity Scale [FSS], Fatigue Scale for Motor and Cognitive Functions [FSMC], Post-Exertional Malaise questionnaire [PEM]), sleep quality (Pittsburgh Sleep Quality Index [PSQI]), daytime sleepiness (Epworth Sleepiness Scale [ESS]), functioning (Sheehan Disability Scale [SDS]), anxiety (Beck Anxiety Inventory [BAI]) and an exploratory adverse effect screening. Follow-up assessments will be performed three days after treatment completion and again at three months post-intervention to evaluate both short- and medium-term effects. Biospecimen collection will include approximately 141 ml of peripheral blood per participant across three time points (baseline, post-treatment, +3 days). Samples will be analyzed for inflammatory markers and securely stored in the institutional biobank of the Max Planck Institute of Psychiatry in accordance with data protection and ethical guidelines. Safety and tolerability will be continuously monitored, including documentation of adverse events. The results of this pilot study are expected to provide preliminary evidence on whether accelerated iTBS protocols may exert differential effects on neuroinflammatory processes and depressive symptomatology in patients with Post-COVID-19 condition, thereby informing larger controlled clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Capacity to consent (legally competent, written informed consent including data protection)
* Diagnosis of depression (at least moderate severity, BDI-II ≥ 20), including major depressive episode in bipolar disorder
* Comorbid diagnosis of Post-COVID-19 condition (WHO definition)
* Insufficient improvement of depressive symptoms under psychopharmacological treatment
* Stable psychopharmacological medication for at least 4 weeks prior to start of iTBS

Exclusion Criteria:

* Age <18 years or >65 years
* Pregnancy, planned pregnancy, or breastfeeding
* Legal guardianship or cognitive impairment preventing valid informed consent
* Severe developmental disorder or intellectual disability
* Acute or chronic substance abuse (alcohol, prescription drugs, or illicit drugs)
* Current treatment with benzodiazepines or Z-substances
* Acute suicidality
* Psychotic symptoms
* Severe neurological disorder (e.g., major brain injury, neurodegenerative disease)
* Ongoing treatment with another neurostimulation method (ECT, TMS, VNS)
* Contraindications to TMS, including: Intracranial metal, implants, shunts, Cochlear implant, pacemaker, implantable defibrillator, History of seizures or epileptiform EEG
* Severe general medical illness (e.g., anemia requiring transfusion, severe arrhythmias, cardiomyopathy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in immunophenotypic marker CRP from baseline to post-treatment | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment
  Differences in CRP from baseline to post-treatment between intensified iTBS and standard iTBS in inflammatory markers (based on material extracted from peripheral blood)
Change in immunophenotypic marker TNF from baseline to post-treatment | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment
  Differences in TNF from baseline to post-treatment between intensified iTBS and standard iTBS in inflammatory markers (based on material extracted from peripheral blood)
Change in immunophenotypic marker IL-1ß from baseline to post-treatment | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment
  Differences in IL-1ß from baseline to post-treatment between intensified iTBS and standard iTBS in inflammatory markers (based on material extracted from peripheral blood)
Change in immunophenotypic marker IL-6 from baseline to post-treatment | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment
  Differences in IL-6 from baseline to post-treatment between intensified iTBS and standard iTBS in inflammatory markers (based on material extracted from peripheral blood)
Total score change in the Becks Depression Inventory, version 2 (BDI-II, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in depression symptomatology, comparison between two arms. Range of the test is 0-63, a higher score indicates a worse condition.
Total score change in the clinician-rated Montgomery Asberg Depression scale (MADRS) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in depression symptomatology, comparison between two arms. Overall score range 0-60, a higher score indicates a more severe depression.

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale (FSS, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in fatigue severity. Comparison between two arms. Overall score range 9-63, higher scores indicate more severe fatigue.
Change in Fatigue Scale for Motor and Cognitive Functions (FSMC, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in fatigue across motor and cognitive domains. Comparison between two arms. Overall score range 20-100, higher scores indicate more severe fatigue.
Change in Post-Exertional Malaise (PEM) Questionnaire (self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in post-exertional malaise symptoms, comparison between arms. Exploratory; no standardized range universally defined.
Change in Pittsburgh Sleep Quality Index (PSQI, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in sleep quality, comparison between arms. Global score range 0-21, higher scores indicate worse sleep quality
Change in Epworth Sleepiness Scale (ESS, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in daytime sleepiness, comparison between arms. Total score range 0-24, higher scores indicate greater daytime sleepiness.
Change in Sheehan Disability Scale (SDS, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in functional impairment across work/school, social, and family life. Each domain scored 0-10; higher scores indicate greater impairment, comparison between arms.
Change in Beck Anxiety Inventory (BAI, self-rating) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Change in self-rated anxiety severity. Total score range 0-63, higher scores indicate more severe anxiety. Comparison between arms.
Adverse Event Screening (Exploratory) | baseline (day of first treatment), day of 15th treatment, 3 days after 30th (last) treatment, follow-up 3 months after treatment completion
  Incidence of adverse events related to iTBS treatment: headache, scalp discomfort, dizziness, sleepiness, fatigue, and other stimulation-related complaints

CONTACTS AND LOCATIONS:
Overall Officials: Angelika Erhardt-Lehmann, MD, Prof., Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max-Planck-Institute of Psychiatry, Munich, Bavaria, Germany